CLINICAL TRIAL: NCT03859947
Title: Comparison of Heated humidiﬁed High-flow Nasal Cannula Flow Rates (1-L/kg/Min vs 2-L/kg/Min) in the Management of Severe Bronchiolitis
Brief Title: High-flow Nasal Cannula Flow Rates, Severe Bronchiolitis
Status: Completed | Type: Observational
Sponsor: Ali Yurtseven (Other)
Collaborators: Ege University (Other)
Responsible Party: Sponsor-Investigator, Ali Yurtseven, Principal Investigator, Ege University
Organization: Ege University (Other)
Other Study IDs: 2.100.2017.0025
Record Dates: First submitted 2019-02-25; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Non-invasive Ventilation; Pediatric Pulmonary Disease
Keywords: Bronchiolitis; Emergency department; High-flow nasal cannula; Flow rate
MeSH Terms: conditions — Bronchiolitis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute bronchiolitis
  Interventions: Device: Heated humidiﬁed high-flow nasal cannula

INTERVENTIONS:
Device: Heated humidiﬁed high-flow nasal cannula — Non-invasive ventilation with a nasal cannula

SUMMARY:
Objective: The investigators aimed to compare the heated humidified high-ﬂow nasal cannula (HHHFNC) flow rate of 1-L/kg/min (1L) with 2-L/kg/min (2L) in patients with severe bronchiolitis presenting to the pediatric emergency department.

Study design: The investigators performed a study in which all patients were allocated to receive these two flow rates. The primary outcome was admitted as treatment failure, which was defined as a clinical escalation in respiratory status. Secondary outcomes covered a decrease of respiratory rate (RR), heart rate (HR), the clinical respiratory score (CRS), rise of peripheral capillary oxygen saturation (SpO2) and rates of weaning, intubation and intensive care unit (ICU) admission.

Keywords: Bronchiolitis, Emergency department, High-flow nasal cannula, Flow rate

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe bronchiolitis
* Must be less than 24 months
* Must have presented to the emergency department

Exclusion Criteria:

* Immediate invasive ventilation and/or intensive care unit admission
* Congenital heart disease,
* Chronic lung disease
* Neuromuscular disease
* Netabolic disease
* Craniofacial anomalies
* Immunocompromised
* Bacterial pneumonia
* Pneumothorax
* Nasal trauma

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All patients with a clinical diagnosis of severe bronchiolitis, aged less than 24 months and presenting to the emergency department
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Treatment failure rate | Within 24 hours
  We compared the treatment failure between the 1-L/kg/min flow rate with 2-L/kg/min rate in patients with severe bronchiolitis

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University School of Medicine, Pediatric Emergency Department, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided